CLINICAL TRIAL: NCT00750581
Title: An Escalating Dose Indomethacin for the Treatment of Persistent Patent Ductus Arteriosus (PDA) In Preterm Infants- A Randomized Pilot Study
Brief Title: An Escalating Dose Indomethacin for the Treatment of Persistent Patent Ductus Arteriosus (PDA) In Preterm Infants
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study medication was no longer available for study
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Amuchou Soraisham, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RT734510
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose group (Placebo Comparator): The infants randomized to the standard dose group will receive indomethacin (0.1 mg/kg) at 24 hr intervals for 5 days. These infants will also receive 5 extra doses of normal saline infusion of similar volume at 12 hrly intervals between the indomethacin schedules to match the Escalating dose Indomethacin Schedule
  Interventions: Drug: Indomethacin
- Escalating dose group (Active Comparator): The infants randomized to the Escalating dose group will receive indomethacin started at 0.2 mg/kg/dose every 12 hours for 2 doses with stepwise increment in indomethacin dose by 0.1 mg/kg/dose every 24 hours upto maximum dose of 0.6 mg/kg/dose
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Indomethacin — Infants randomized to Escalating Dose group will receive indomethacin (0.2 mg/kg/dose) at 12 hr intervals for 2 doses, followed by indomethacin (0.3 mg/kg/dose) at 12 hr interval for 2 doses, then Indomethacin (0.4 mg/kg/dose) at 12 hr interval for 2 doses, increased to indomethacin (0.5 mg/kg/dose) at 12 hour interval for 2 doses and finally indomethacin 0.6 mg/kg/dose at 12 hourly interval for 2 doses.
  Other Names: indocid

SUMMARY:
A large patent ductus arteriosus (PDA) is associated with congestive heart failure, pulmonary hemorrhage, chronic lung disease (CLD), necrotizing enterocolitis (NEC) and intraventricular bleeding. Indomethacin is the first line of treatment for PDA. Failure of ductal closure with the first course of indomethacin is reported in 30-40% of infants, with a higher failure rate in infants weighing < 1000 gm. PDA ligation is associated with early postoperative hypotension, oxygenation failure and adverse neurodevelopmental outcome in preterm infants. The use of escalating doses of Indomethacin in the treatment of persistent PDA was found to be safe and decreased the need for PDA ligation without adverse effects in one observational study.We hypothesize that the use of an escalated dose of intravenous indomethacin will result in an increase in the probability of survival without need for surgical ligation of PDA as compared to a standard dose indomethacin in newborn infants < 29 weeks of gestational age with persistent PDA.

DETAILED DESCRIPTION:
This study is a randomized control trial.Those eligible infants will be randomized to either a Standard Dose group or to Escalating Dose indomethacin group after obtaining parental consent. The infants randomized to the standard dose group will receive indomethacin (0.1 mg/kg) at 24 hr intervals for 5 days. Escalating Dose group infants will receive indomethacin (0.2 mg/kg/dose) at 12 hr intervals for 2 doses, followed by indomethacin (0.3 mg/kg/dose) at 12 hr interval for 2 doses, then Indomethacin (0.4 mg/kg/dose) at 12 hr interval for 2 doses, increased to indomethacin (0.5 mg/kg/dose) at 12 hour interval for 2 doses and finally indomethacin 0.6 mg/kg/dose at 12 hourly interval for 2 doses. To keep the study blinded, the standard group will receive 5 extra doses of normal saline infusion of similar volume at 12 hrly intervals between the indomethacin schedules to match the Escalating dose Indomethacin Schedule. Daily Echo will be performed and if the Echo showed closure of PDA after 3 days of assigned treatment, no further indomethacin will be given in both the groups.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age < 29 weeks and/or birth weight < 1251gm
* Presence of PDA after completion of first course of indomethacin

Exclusion Criteria:

* Infants with PDA dependent congenital heart disease
* Chromosomal or major congenital anomalies
* Infants in whom use of indomethacin is contraindicated.(i.e.infants with acute renal failure,necrotizing enterocolitis,severe thrombocytopenia (platelet count < 60,000/ mm3) and evidence of clinical bleeding (pulmonary bleeding, severe intraventricular bleeding grade 3&4)

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Survival without PDA ligation at discharge | till the discharge from hospital

SECONDARY OUTCOMES:
PDA closure rate | after completion of indomethacin treatment
Incidence of necrotizing enterocolitis, renal failure and bronchopulmonary dysplasia | till discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Amuchou S Soraisham, MD, DM, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada